CLINICAL TRIAL: NCT03618719
Title: Impact of Intermittent Hypoxia on Phagocytosis and Sepsis Outcomes: the Potential Role of Statin (Part III: Human Study in 2018-2019)
Brief Title: Impact of Intermittent Hypoxia on the Function of the Phagocytes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016-06-005CC
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: obstructive sleep apnea; intermittent hypoxia; granulocyte function; continuous positive airway pressure (CPAP) therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — white cells in peripheral venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obstructive sleep apnea: Patients with treatment-naive obstructive sleep apnea (OSA) who need continuous positive airway pressure (CPAP) therapy on clinical basis
- Control: Healthy controls without OSA

SUMMARY:
Patients with treatment-naive obstructive sleep apnea (OSA) who need continuous positive airway pressure (CPAP) therapy on clinical basis are included as well as healthy controls without OSA. 15 cc peripheral venous blood is drawn on the date of diagnosis of OSA and 3-6 months after CPAP therapy. Granulocytes are harvested and tested for its function, such as phagocytosis, reactive oxygen species (ROS) production and bacteria-killing ability.

DETAILED DESCRIPTION:
Patients with treatment-naive obstructive sleep apnea (OSA) who need continuous positive airway pressure (CPAP) therapy on clinical basis are included. Healthy controls without OSA are enrolled, too. 15 cc peripheral venous blood is drawn on the date of diagnosis of OSA and 3-6 months after CPAP therapy (not given to controls). Granulocytes are harvested and tested for its function, such as phagocytosis, reactive oxygen species (ROS) production and bacteria-killing ability.

ELIGIBILITY:
Inclusion Criteria:

<OSA group> 1. Patients with treatment-naive obstructive sleep apnea (OSA) who need continuous positive airway pressure (CPAP) therapy on clinical basis 2. aged 20 years or older 3. Apnea-hypopnea index (AHI) at least 15/hour 4. Willing to participate this study <Control group>

1. Healthy controls without OSA
2. aged 20 years or older
3. AHI less than 5/hour

Exclusion Criteria:

<OSA group>

1. OSA patients who do not need continuous positive airway pressure (CPAP) therapy
2. OSA Patients have ever received CPAP or other treatment
3. aged less than 20 years
4. AHI at least 15/hour
5. Not willing to participate this study <Control group>

1. Apnea-hypopnea index (AHI) equals to or more than 5/hour 2. aged less than 20 years 3. Not willing to participate this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: <OSA group> Adult Patients with treatment-naive obstructive sleep apnea (OSA) who need continuous positive airway pressure (CPAP) therapy on clinical basis are included.
  <Control group> Healthy adult controls without OSA
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-07-03 (Estimated); Study Completion 2019-07-03 (Estimated)

PRIMARY OUTCOMES:
Granuolocyte function | On enrollment
  Granuolocyte function, such as such as phagocytosis, reactive oxygen species (ROS) production and bacteria-killing ability.
Granuolocyte function | 3-month
  Granuolocyte function, such as such as phagocytosis, reactive oxygen species (ROS) production and bacteria-killing ability.
Granuolocyte function | 6-month
  Granuolocyte function, such as such as phagocytosis, reactive oxygen species (ROS)

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ta Chou, M.D, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Chest department, Taipei Veteran General Hospital, Taipei, Taiwan